CLINICAL TRIAL: NCT06366165
Title: The Effect of Using Seemingly Irrelevant Videos and Memes in Teaching Special Care Dentistry Curriculum
Brief Title: Linking Special Care Dentistry Curriculum to Seemingly Irrelevant Comedy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ACU-Med3
Record Dates: First submitted 2024-04-07; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Learning Problem
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Testing the procedure of using a different mode of teaching medical content
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Students of semester 9 in Ahram Canadian University (Experimental): The students receive their lectures with funny videos and memes included to link the science with it.
  Interventions: Procedure: seemingly irrelevant funny videos and memes in teaching

INTERVENTIONS:
Procedure: seemingly irrelevant funny videos and memes in teaching — linking funny videos and memes to special care dentistry curriculum lectures

SUMMARY:
As Special care dentistry curriculum is very complicated and has a lot of details. Upon teaching it, the investigator will include memes and videos of movies and cartoons and will test the degree of retention of the information after years of passing the subject's exam.

ELIGIBILITY:
Inclusion Criteria:

* students in Ahram Canadian University.
* students who passed Special care dentistry course.
* students who were enrolled in the course from Fall 2021 to Summer 2023

Exclusion Criteria:

* Students who refused to answer the questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
degree of retention of information | from 1 to 3 years
  online questionnaire sent to graduates

CONTACTS AND LOCATIONS:
Locations (1):
- Ahram Candian University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No